CLINICAL TRIAL: NCT06256432
Title: A Multi-Centre, Randomised, Open-Label, Phase II Study of Ambrisentan in Patients With Hepatorenal Syndrome
Brief Title: Endothelin Receptor Antagonism With Ambrisentan to Treat Hepatorenal Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Noorik Biopharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-003-CRD005
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Hepatorenal Syndrome; Liver Cirrhosis; Acute Kidney Injury; Ascites Hepatic
MeSH Terms: conditions — Hepatorenal Syndrome; Liver Cirrhosis; Acute Kidney Injury | interventions — ambrisentan; Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ambrisentan - Low Dose 1 (Experimental): Liquid solution for oral administration, dose < 250 µg/day, up to 60 days
  Interventions: Drug: Ambrisentan
- Ambrisentan - Low Dose 2 (Experimental): Liquid solution for oral administration, dose < 250 µg/day, up to 60 days
  Interventions: Drug: Ambrisentan
- Terlipressin (Active Comparator): Sterile lyophilized powder, to be reconstituted for intravenous administration, at a dose indicated by the study investigator and administered for up to 14 days, considering the following recommendation: 1 mg terlipressin administered in 2-minute bolus every 6 hours for 3 days, and dose of terlipressin increased to 2 mg every 6 hours in the absence of a decrease of at least 30% in serum creatinine by day 4
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Ambrisentan — Endothelin receptor antagonist
  Arms: Ambrisentan - Low Dose 1; Ambrisentan - Low Dose 2
Drug: Terlipressin — Terlipressin
  Arms: Terlipressin

SUMMARY:
Patients with advanced cirrhosis of the liver develop kidney problems occasionally. This condition is called Hepatorenal Syndrome, requires hospitalization and frequently results in death.

The goal of this clinical trial is to test whether the administration of low doses of ambrisentan can help patients with Hepatorenal Syndrome and to determine if it is safe. Ambrisentan is a drug that is approved for the treatment of high blood pressure in the lungs at higher doses.

This clinical trial will compare the safety and effects of ambrisentan to another drug called terlipressin, which is commonly used to treat patients with hepatorenal syndrome.

The main questions the clinical trial aims to answer are:

* Does ambrisentan help the kidney function of the patient?
* Does ambrisentan help prevent death in patients with Hepatorenal Syndrome?
* Does ambrisentan prevent Hepatorenal Syndrome from reappearing?

While in the hospital, trial participants will receive either one of two doses of ambrisentan or terlipressin. If in the first 4 days, ambrisentan is not helpful, the patient may be eligible to receive terlipressin. Patients assigned to receive ambrisentan will continue taking this medication at home after leaving the hospitals and until they complete 60 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent prior to any study-related procedures.
* Age ≥ 18 years and ≤ 70 years.
* Male or non-pregnant, non-lactating female. Women of child-bearing potential must have a confirmed negative serum pregnancy test at the time of screening and must use a highly effective contraceptive method throughout the study such as combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tube occlusion, vasectomised partner, and sexual abstinence and until one month after completing treatment with the study medication. In the case of hormonal contraception, women should have been on a stable regimen for a minimum of three months before study enrolment. Women not of child-bearing potential include post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy). Men must use an effective contraception method (i.e., condom + diaphragm/spermicidal gel or foam, or vasectomy), and should not donate semen during the study. Men are considered to be fertile from the time of puberty, except for those men with permanent sterility secondary to bilateral orchiectomy.
* Cirrhosis of the liver by laboratory examination, clinical history or biopsy.
* History of ascites.
* Increase in serum creatinine ≥ 0.3 mg/dl (26.5 µmol/L) from a value obtained in the 7 days prior to admission, OR a serum creatinine ≥ 1.5 mg/dl (132.6 µmol/L) and is ≥ 1.5-fold above the most recent and lowest value obtained in the last 3 months.
* The subject has no clinical and/or haemodynamic evidence of intravascular volume depletion; or has undergone at least 12 hours of diuretic withdrawal and fluid resuscitation to discard or treat intravascular volume depletion (such as difficulty in establishing volume status, volume status is assessed as equivocal, or there is clinical and/or haemodynamic evidence of intravascular volume depletion), and no significant improvement in serum creatinine has been observed.

Exclusion Criteria:

* Serum creatinine > 5 mg/dL (442 µmol/L).
* Mean arterial pressure (MAP) < 60 mmHg.
* Large Volume Paracentesis (LVP) in the 3 days prior to screening.
* Sepsis, uncontrolled bacterial infection or less than 2 days anti-infective therapy for documented or suspected bacterial infection.
* Total bilirubin > 8 mg/dL (137 µmol/L).
* Serum sodium < 125 mmol/L.
* International Normalised Ratio (INR) ≥ 3.5.
* Proteinuria ≥ 1000 mg/dL.
* Microhaematuria > 50 red blood cells per high power field.
* Clinically significant casts on urinalysis, including granular casts.
* History or evidence of obstructive uropathy or parenchymal renal disease on ultrasound or other imaging.
* Subject with a recent history of circulatory shock defined as MAP < 60 mmHg within 5 days prior to screening requiring vasopressors or subjects requires circulatory support with vasopressors during screening.
* Subject requiring oxygen supplementation or mechanical ventilation.
* Recent exposure to nephrotoxic agents or exposure to radiographic contrast agents within 72 hrs prior to screening.
* Superimposed acute liver failure/injury due to factors other than alcohol, including acute viral hepatitis, drugs, medications (e.g., acetaminophen), or other toxins (e.g., mushroom [Amanita] poisoning).
* Severe cardiovascular disease, including, but not limited to, unstable angina, pulmonary oedema, congestive heart failure (NYHA ≥ II), or persisting symptomatic peripheral vascular disease, myocardial infarction or stable chronic angina within the past 12 months, or any other cardiovascular disease judged by the Investigator to be severe.
* Subject has a history of Transjugular Intrahepatic Portosystemic shunt (TIPS).
* Subject with acute variceal bleeding at the time of screening who may undergo pre-emptive TIPS or is anticipated to be treated with terlipressin.
* Current or recent Renal Replacement Therapy (RRT) within 30 days of enrolment, or anticipation of RRT in the next 3 days after screening.
* Hepatocellular Carcinoma (HCC) beyond the Milan criteria or other malignancy affecting survival beyond 6 months.
* Participation in a study of an investigational medical product or device within the last 30 days preceding screening.
* Hepatic Encephalopathy with West Haven Grade III or IV.
* Current or recent (30 days prior to enrolment) treatment with endothelin receptor antagonists, including ambrisentan.
* Estimated life expectancy of less than 3 days.
* Known allergy or sensitivity to ambrisentan or propylene glycol.
* History of Idiopathic Pulmonary Fibrosis.
* Subject is unable or unwilling to follow instructions or comply with study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in estimated GFR (eGFR) from baseline | 4 days
  As determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula

SECONDARY OUTCOMES:
Proportion of patients achieving Hepatorenal Syndrome reversal | 14 days
  Reversal defined as two consecutive serum creatinine values < 1.5 mg/dL (132 µmol/L) within 24 hours
Proportion of subjects experiencing Hepatorenal Syndrome recurrence | 60 days
  Recurrence defined as the appearance of Hepatorenal Syndrome satisfying all clinical trial entry criteria
Overall survival | 60 days
  Proportion of participants alive in each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Iker Navarro, MD, Study Director — Noorik Biopharmaceuticals AG
Locations (6):
- India (6):
  - Aster CMI Hospital, Bangalore, Karnataka
  - Sir HN Reliance Hospital Foundation, Mumbai, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Asian Institute of Gastroenterology (AIG), Hyderabad, Telangana
  - Ganesh Shankar Vidyarthi Memorial (GSVM) Medical College, Kanpur, Uttar Pradesh
  - Medanta Multi Super Specialty Hospital, Lucknow, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Angeli P, Gines P, Wong F, Bernardi M, Boyer TD, Gerbes A, Moreau R, Jalan R, Sarin SK, Piano S, Moore K, Lee SS, Durand F, Salerno F, Caraceni P, Kim WR, Arroyo V, Garcia-Tsao G; International Club of Ascites. Diagnosis and management of acute kidney injury in patients with cirrhosis: revised consensus recommendations of the International Club of Ascites. Gut. 2015 Apr;64(4):531-7. doi: 10.1136/gutjnl-2014-308874. Epub 2015 Jan 28. No abstract available. PMID 25631669
- [Background] Soper CP, Latif AB, Bending MR. Amelioration of hepatorenal syndrome with selective endothelin-A antagonist. Lancet. 1996 Jun 29;347(9018):1842-3. No abstract available. PMID 8667963
- [Background] Mindikoglu AL, Weir MR. Current concepts in the diagnosis and classification of renal dysfunction in cirrhosis. Am J Nephrol. 2013;38(4):345-54. doi: 10.1159/000355540. Epub 2013 Oct 5. PMID 24107793
- [Background] Ring-Larsen H. Renal blood flow in cirrhosis: relation to systemic and portal haemodynamics and liver function. Scand J Clin Lab Invest. 1977 Nov;37(7):635-42. doi: 10.3109/00365517709100657. PMID 594643
- [Background] Moore K. Endothelin and vascular function in liver disease. Gut. 2004 Feb;53(2):159-61. doi: 10.1136/gut.2003.024703. PMID 14724140
- [Background] Moore K, Wendon J, Frazer M, Karani J, Williams R, Badr K. Plasma endothelin immunoreactivity in liver disease and the hepatorenal syndrome. N Engl J Med. 1992 Dec 17;327(25):1774-8. doi: 10.1056/NEJM199212173272502. PMID 1435931
- [Background] Zipprich A, Gittinger F, Winkler M, Dollinger MM, Ripoll C. Effect of ET-A blockade on portal pressure and hepatic arterial perfusion in patients with cirrhosis: A proof of concept study. Liver Int. 2021 Mar;41(3):554-561. doi: 10.1111/liv.14757. Epub 2021 Jan 5. PMID 33295121
- [Background] Dhaun N, Macintyre IM, Melville V, Lilitkarntakul P, Johnston NR, Goddard J, Webb DJ. Blood pressure-independent reduction in proteinuria and arterial stiffness after acute endothelin-a receptor antagonism in chronic kidney disease. Hypertension. 2009 Jul;54(1):113-9. doi: 10.1161/HYPERTENSIONAHA.109.132670. Epub 2009 Jun 8. PMID 19506099
- [Background] Wong F, Moore K, Dingemanse J, Jalan R. Lack of renal improvement with nonselective endothelin antagonism with tezosentan in type 2 hepatorenal syndrome. Hepatology. 2008 Jan;47(1):160-8. doi: 10.1002/hep.21940. PMID 17886336